CLINICAL TRIAL: NCT06146634
Title: Washington State Driving Intervention Research Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Academy of Sciences (Unknown); The Driver Training Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00025991
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Driving Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hazard Perception Training (Experimental)
  Interventions: Behavioral: Hazard Perception Training
- Vehicle Maintenance Training (Placebo Comparator)
  Interventions: Behavioral: Vehicle Maintenance Training
- Attention Maintenance Training (Active Comparator)
  Interventions: Behavioral: Attention Maintenance Training
- ZED Training (No Intervention)

INTERVENTIONS:
Behavioral: Hazard Perception Training — The hazard perception training is comprised of three modules. Each module is comprised of four scenarios. Each hazard perception scenario has two activities. The entire training is expected to take approximately an hour to complete.
  Arms: Hazard Perception Training
Behavioral: Vehicle Maintenance Training — For participants randomized into the placebo group, they will receive a brief training on vehicle maintenance using a series of short videos. These videos describe regular checks that drivers should do, such as checking windshield wiper fluid levels, and how to change engine oil. Altogether the videos will last approximately 1 hour.
  Arms: Vehicle Maintenance Training
Behavioral: Attention Maintenance Training — The attention maintenance training is comprised of three modules. Each module is comprised of four scenarios, with each scenario corresponding to one activity. The entire training is expected to take approximately an hour to complete.
  Arms: Attention Maintenance Training

SUMMARY:
The goal of this clinical trial is to test the effect of hazard perception and attention maintenance training and testing on driving performance. Participants will be randomized into a treatment group receiving hazard perception or attention maintenance training or a control group receiving either vehicle maintenance training or the status quo ZED training. Randomization will occur by location. Researchers will compare the treatment and control groups to see if there are differences in driving behavior and crash rates.

DETAILED DESCRIPTION:
The experiment's purpose is to assess the performance of the investigator's novel Driving Hazard Perception and Attention Maintenance training intervention on improving related driving skills, performance in driving exams, and long-term benefits as assessed by crash statistics and naturalistic driving behavior. A two-group pre-post experimental design will be used to evaluate the effectiveness of the new Driving Hazard Perception Training. Each training (hazard perception and attention maintenance) will be assessed in relation to the status quo (ZED training) and in relation to a placebo that has no training related to hazard perception or attention maintenance (vehicle maintenance training). Participants beginning a driver education program will be recruited. Each participating location will be randomized to one of the four research arms. Baseline hazard perception assessment will be performed first, and then participants will receive one of the four trainings. Lastly, all participants will take a hazard perception exam to assess the participants' performance. All participants will also use a smartphone application to collect driving data during the learner driver period and 12 months of independent driving. Driving behaviors and state-level crash data will be used to assess the impact of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a driver training course through the 911 driving school in Washington State.

Exclusion Criteria:

* Participants must meet the above criteria.
* Additionally, participants will be excluded if either the participant or the participant's parent opts-out.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Crashes | Post-licensure up to 12 months
  The number of participant-involved crashes.
Number of Near-crashes | Post-licensure up to 12 months
  The number of participant-involved near-crashes.
Longitudinal g-force events | Post-licensure up to 12 months
  Significant longitudinal g-force events greater than 0.5 g
Lateral g-force events | Post-licensure up to 12 months
  Significant lateral g-force events greater than 0.5 g

CONTACTS AND LOCATIONS:
Overall Officials: Johnathon Ehsani, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- The Driver Training Group, Seattle, Washington, United States